CLINICAL TRIAL: NCT03214029
Title: COmparisoN of High-sensitivity Cardiac TRoponin I and T ASsays Trial
Acronym: CONTRAST
Status: Active, not recruiting | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Abbott Diagnostics Division (Industry); Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Sponsor
Other Study IDs: CONTRAST
Record Dates: First submitted 2017-06-26; First posted 2017-07-11 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Acute Myocardial Infarction; Acute Coronary Syndrome
Keywords: troponin; high-sensitivity cardiac troponin; acute myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Excess blood is biobanked as EDTA-plasma and heparin samples after being used for the clinical cTnI assay
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Study population: Prospective, observational cohort study of consecutives patients (goal, 2000 patients over 5 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
  Interventions: Diagnostic Test: Cardiac troponin testing

INTERVENTIONS:
Diagnostic Test: Cardiac troponin testing — Fresh EDTA plasma samples will be measured with both the hs-cTnI (Abbott) and hs-cTnT (Roche) assays.

SUMMARY:
Compare the analytical and clinical performance of hs-cTnI and hs-cTnT assays for the diagnosis of acute myocardial injury and myocardial infarction in patients presenting to the emergency department in whom serial cTnI measurements are obtained on clinical indication.

DETAILED DESCRIPTION:
Background: Comparative studies addressing the analytical and clinical performance of hs-cTnI and hs-cTnT assays for the diagnosis of acute myocardial injury and myocardial infarction in consecutive patients presenting to a United States (US) emergency department are lacking.

Study objective: Compare the analytical and clinical performance of hs-cTnI and hs-cTnT assays for the diagnosis of acute myocardial injury and myocardial infarction in patients presenting to the emergency department in whom serial cTnI measurements are obtained on clinical indication.

Null Hypothesis: hs-cTnI and or hs-cTnT assays will offer comparable diagnostic performance for acute myocardial injury and acute myocardial

ELIGIBILITY:
Inclusion Criteria:

1. Adult, defined as subject 18 years of age or older
2. Baseline cTn measurement and at least one additional cTn measurement within 6 hours after initial cTnI measurement.
3. At least one 12-lead electrocardiogram

Exclusion Criteria:

1. Currently pregnant
2. Trauma related admission
3. Cardiac arrest
4. Decline to participate
5. Did not present through the ED
6. Transferred from an outside hospital

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients (goal, 2000 patients over 5 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic outcome analytical comparison of high-sensitivity cardiac troponin I and T assays for the diagnosis of acute myocardial injury and infarction. | on admission
  Diagnostic performance of cardiac troponin assays for the diagnosis of acute myocardial injury and myocardial infarction

SECONDARY OUTCOMES:
All-cause mortality | Up to 180-days
  Any death
Cardiac death | Up to 180-days
  Death due to cardiac reasons.
Unstable angina | Up to 180-days
  Diagnosis of unstable angina per chart review up to 180-days
Acute myocardial infarction | Up to 180-days
  Diagnosis of Acute myocardial infarction per chart review up to 180 days.
Revascularization | Up to 180-days
  Coronary artery bypass graft surgery or percutaneous coronary intervention
Safety outcome: Major adverse cardiac events: cardiac death, unstable angina, acute myocardial infarction, revascularization, and congestive heart failure. | 30-days
  Safety outcome for tested diagnostic strategies will be defined at 30-days, including index hospitalization events for MACE - Major adverse cardiac events: cardiac death, unstable angina, acute myocardial infarction, revascularization, and congestive heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Fred S Apple, PhD, Principal Investigator — Hennepin County Medical Center and Minneapolis Medical Research Foundation
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States